CLINICAL TRIAL: NCT00925171
Title: The Effects of Maintenance Schedules Following Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Maintenance Schedules Following Pulmonary Rehabilitation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Andrew Wilson, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009RESP05; 09/H0304/40
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation; Chronic Respiratory Questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): Intervention with exercise management
  Interventions: Behavioral: Pulmonary Intervention
- Control Group (No Intervention): Patients will receive the standard advice to undertake strength and endurance exercises at home and invitation to attend the Norwich Breath Easy Group
  Patients will be stratified according to whether the initial programme took place in the outpatient hospital or community setting

INTERVENTIONS:
Behavioral: Pulmonary Intervention — Maintenance programme of 2 hours duration, every 3 months. During the first hour patients will describe the extent to which they have been able to continue with their exercises at home on an individual basis and ways of enhancing adherence to this training will be discussed. Positive re-enforcement will be provided. Patients with suspected depression or social isolation will be referred to their GP for additional management. Patients will be advised on dyspnoea management strategies, especially controlled breathing combined with supervised activity exertion on activities relevant to their daily living. This will be followed by 1 hour of supervised strength and endurance training including walking, cycling, standing from sitting, arm exercises using dumbbells and step-ups. Patients will receive a written report on their progress by their physician and copied to their GP. This will be in addition to the standard advice given to the control group.
  Arms: Pulmonary Rehabilitation Group

SUMMARY:
Chronic obstructive pulmonary disease (COPD), a preventable and treatable condition, is a major healthcare problem with huge human and economic costs. It affects 3 million people, results in 1.4 million consultations, causes 30,000 deaths, and costs £800M per year in the UK. Considerable research expenditure is devoted to finding new and expensive interventions. However pulmonary rehabilitation (PR) is an available therapeutic option with good evidence of benefit for patients in terms of quality of life and daily functioning.

The primary objective of the study is to evaluate the effectiveness and cost effectiveness of the addition of a maintenance programme following pulmonary rehabilitation in patients with COPD when compared to standard care.

The secondary objective is to identify baseline characteristics that will predict improvement in pulmonary rehabilitation programmes and adherence to maintenance strategies. By measuring a series of demographic, clinical, physiological, psychological and biochemical parameters the researchers hope to be able to predict those patients who are likely to receive the greatest benefit from pulmonary rehabilitation.

An additional objective will be to prepare a detailed maintenance programme manual. This will be available to other centres providing pulmonary rehabilitation at the conclusion of the study

DETAILED DESCRIPTION:
This will be a randomised, controlled, parallel study of a maintenance pulmonary rehabilitation (PR) programme in patients with chronic obstructive pulmonary disease (COPD). Following successful completion of a PR programme in Norwich(see below) patients will be randomised to receive maintenance PR or standard medical care.

Prior to enrolment in the PR programme, patients will undergo standard baseline assessments, after providing informed consent. These will include a medical examination, demographic details, past medical history, spirometry, an incremental shuttle walk test (ISWT) to determine a predicted maximum oxygen consumption, an endurance shuttle walk test (ESWT) at 85% of predicted maximum oxygen consumption (V02), chronic respiratory questionnaire (CRQ), EuroQol (EQ5D), hospital anxiety and depression score (HADS), serum interleukin(IL)-6 and C-reactive protein (CRP), body mass index (BMI), skinfold thickness and muscle strength.

At the end of PR and twelve months following PR patients will undergo medical examination, ESWT at 85% of predicted maximum VO2, CRQ, EQ5D, HADS, serum interleukin(IL)-6 and CRP, BMI, skinfold thickness and muscle strength and an assessment of activity in the preceding month.

At 3 months, 6 months and 9 months following PR patients will complete the CRQ and a questionnaire to assess activity in the preceding month. These will be undertaken by postal questionnaire.

Baseline socioeconomic and costs questionnaire will be completed at entry to the PR and follow-up cost questionnaires will be completed following PR and after 3, 6, 9 and 12 months. Patients will be given a diary card on which to record NHS contacts, prescriptions etc at all visits.

The 3, 6 and 9-month questionnaires will be collected by post.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 35 years
* Physician labelled diagnosis of COPD, emphysema or chronic bronchitis
* Ex or current smoker of more than 20 pack years
* FEV1 less than 80% of predicted
* Patients may be taking long or short acting bronchodilators and/or inhaled or oral corticosteroids and/or theophyllines.
* Patients having attended at least 60% of the exercise sessions in the initial PR(22)* * This is an inclusion criterion for randomisation to receive maintenance PR or standard medical care but not entry into the study

Exclusion Criteria:

* Significant cardiac or pulmonary disease other than COPD such that COPD is the minor contribution to the patients' symptoms.
* Myocardial infarction within the previous 6 months or unstable angina
* Respiratory infection defined as cough, antibiotic use or purulent sputum within 4 weeks prior to randomisation.
* Severe or uncontrolled co-morbid disease, which is likely to affect the outcome of the study.
* Abnormalities in cognitive functioning that would limit the patient's ability to undertake the procedures required in the study.
* Unable to give written informed consent.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be change from baseline in the dyspnoea domain of the Chronic Respiratory Questionnaire (CRQ). | 14 Months

SECONDARY OUTCOMES:
Endurance shuttle walk test | 14 months
Fat free mass | 14 Months
Body mass index | 14 Months
Quality Adjusted Life Years (QALY) gained (estimated from EQ-5D data) | 14 Months
Hospital anxiety and depression score (HADS) | 14 Months
Changes in medication and NHS Resource Utilisation including hospitalisations, health professional contact, medication and adverse events | 14 Months
Change in peripheral blood C-reactive protein, Tumour Necrosis Factor (TNF) alpha, Interleukin (IL) 6 | 14 Months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilson, MD MRCP (UK), Principal Investigator — Clinical Senior Lecturer, University of East Anglia
Locations (2):
- United Kingdom (2):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - University of East Anglia, Norwich, Norfolk

REFERENCES:
- [Background] Lacasse Y, Martin S, Lasserson TJ, Goldstein RS. Meta-analysis of respiratory rehabilitation in chronic obstructive pulmonary disease. A Cochrane systematic review. Eura Medicophys. 2007 Dec;43(4):475-85. PMID 18084170
- [Background] Singh SJ, Smith DL, Hyland ME, Morgan MD. A short outpatient pulmonary rehabilitation programme: immediate and longer-term effects on exercise performance and quality of life. Respir Med. 1998 Sep;92(9):1146-54. doi: 10.1016/s0954-6111(98)90410-3. PMID 9926171
- [Background] Ries AL, Bauldoff GS, Carlin BW, Casaburi R, Emery CF, Mahler DA, Make B, Rochester CL, Zuwallack R, Herrerias C. Pulmonary Rehabilitation: Joint ACCP/AACVPR Evidence-Based Clinical Practice Guidelines. Chest. 2007 May;131(5 Suppl):4S-42S. doi: 10.1378/chest.06-2418. PMID 17494825
- [Background] Romagnoli M, Dell'Orso D, Lorenzi C, Crisafulli E, Costi S, Lugli D, Clini EM. Repeated pulmonary rehabilitation in severe and disabled COPD patients. Respiration. 2006;73(6):769-76. doi: 10.1159/000092953. Epub 2006 Apr 21. PMID 16636528
- [Background] Foglio K, Bianchi L, Ambrosino N. Is it really useful to repeat outpatient pulmonary rehabilitation programs in patients with chronic airway obstruction? A 2-year controlled study. Chest. 2001 Jun;119(6):1696-704. doi: 10.1378/chest.119.6.1696. PMID 11399693
- [Background] Ries AL, Kaplan RM, Myers R, Prewitt LM. Maintenance after pulmonary rehabilitation in chronic lung disease: a randomized trial. Am J Respir Crit Care Med. 2003 Mar 15;167(6):880-8. doi: 10.1164/rccm.200204-318OC. Epub 2002 Dec 27. PMID 12505859
- [Background] Brooks D, Krip B, Mangovski-Alzamora S, Goldstein RS. The effect of postrehabilitation programmes among individuals with chronic obstructive pulmonary disease. Eur Respir J. 2002 Jul;20(1):20-9. doi: 10.1183/09031936.02.01852001. PMID 12166571
- [Background] Hui KP, Hewitt AB. A simple pulmonary rehabilitation program improves health outcomes and reduces hospital utilization in patients with COPD. Chest. 2003 Jul;124(1):94-7. doi: 10.1378/chest.124.1.94. PMID 12853508
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones RW, Wedzicha AJ. Longitudinal trends in exercise capacity and health status after pulmonary rehabilitation in patients with COPD. Respir Med. 2003 Feb;97(2):173-80. doi: 10.1053/rmed.2003.1397. PMID 12587969
- [Background] Norweg AM, Whiteson J, Malgady R, Mola A, Rey M. The effectiveness of different combinations of pulmonary rehabilitation program components: a randomized controlled trial. Chest. 2005 Aug;128(2):663-72. doi: 10.1378/chest.128.2.663. PMID 16100152
- [Background] Puente-Maestu L, Sanz ML, Sanz P, Cubillo JM, Mayol J, Casaburi R. Comparison of effects of supervised versus self-monitored training programmes in patients with chronic obstructive pulmonary disease. Eur Respir J. 2000 Mar;15(3):517-25. doi: 10.1034/j.1399-3003.2000.15.15.x. PMID 10759446
- [Background] Sewell L, Singh SJ, Williams JE, Collier R, Morgan MD. Can individualized rehabilitation improve functional independence in elderly patients with COPD? Chest. 2005 Sep;128(3):1194-200. doi: 10.1378/chest.128.3.1194. PMID 16162706
- [Background] Puhan MA, Schunemann HJ, Frey M, Scharplatz M, Bachmann LM. How should COPD patients exercise during respiratory rehabilitation? Comparison of exercise modalities and intensities to treat skeletal muscle dysfunction. Thorax. 2005 May;60(5):367-75. doi: 10.1136/thx.2004.033274. PMID 15860711
- [Background] Arnold E, Bruton A, Ellis-Hill C. Adherence to pulmonary rehabilitation: A qualitative study. Respir Med. 2006 Oct;100(10):1716-23. doi: 10.1016/j.rmed.2006.02.007. Epub 2006 Mar 22. PMID 16554147
- [Background] Jette AM, Rooks D, Lachman M, Lin TH, Levenson C, Heislein D, Giorgetti MM, Harris BA. Home-based resistance training: predictors of participation and adherence. Gerontologist. 1998 Aug;38(4):412-21. doi: 10.1093/geront/38.4.412. PMID 9726128
- [Background] Griffiths TL, Phillips CJ, Davies S, Burr ML, Campbell IA. Cost effectiveness of an outpatient multidisciplinary pulmonary rehabilitation programme. Thorax. 2001 Oct;56(10):779-84. doi: 10.1136/thorax.56.10.779. PMID 11562517
- [Background] Redelmeier DA, Guyatt GH, Goldstein RS. Assessing the minimal important difference in symptoms: a comparison of two techniques. J Clin Epidemiol. 1996 Nov;49(11):1215-9. doi: 10.1016/s0895-4356(96)00206-5. PMID 8892486
- [Background] Williams JE, Singh SJ, Sewell L, Morgan MD. Health status measurement: sensitivity of the self-reported Chronic Respiratory Questionnaire (CRQ-SR) in pulmonary rehabilitation. Thorax. 2003 Jun;58(6):515-8. doi: 10.1136/thorax.58.6.515. PMID 12775865
- [Background] de Torres JP, Pinto-Plata V, Ingenito E, Bagley P, Gray A, Berger R, Celli B. Power of outcome measurements to detect clinically significant changes in pulmonary rehabilitation of patients with COPD. Chest. 2002 Apr;121(4):1092-8. doi: 10.1378/chest.121.4.1092. PMID 11948037
- [Background] Moullec G, Ninot G, Varray A, Desplan J, Hayot M, Prefaut C. An innovative maintenance follow-up program after a first inpatient pulmonary rehabilitation. Respir Med. 2008 Apr;102(4):556-66. doi: 10.1016/j.rmed.2007.11.012. Epub 2007 Dec 27. PMID 18164191
- [Background] Berry MJ, Rejeski WJ, Adair NE, Ettinger WH Jr, Zaccaro DJ, Sevick MA. A randomized, controlled trial comparing long-term and short-term exercise in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2003 Jan-Feb;23(1):60-8. doi: 10.1097/00008483-200301000-00011. PMID 12576914
- [Background] Puhan MA, Guyatt GH, Goldstein R, Mador J, McKim D, Stahl E, Griffith L, Schunemann HJ. Relative responsiveness of the Chronic Respiratory Questionnaire, St. Georges Respiratory Questionnaire and four other health-related quality of life instruments for patients with chronic lung disease. Respir Med. 2007 Feb;101(2):308-16. doi: 10.1016/j.rmed.2006.04.023. Epub 2006 Jun 19. PMID 16782320
- [Background] Guyatt GH, Berman LB, Townsend M, Pugsley SO, Chambers LW. A measure of quality of life for clinical trials in chronic lung disease. Thorax. 1987 Oct;42(10):773-8. doi: 10.1136/thx.42.10.773. PMID 3321537
- [Background] Singh SJ, Sodergren SC, Hyland ME, Williams J, Morgan MD. A comparison of three disease-specific and two generic health-status measures to evaluate the outcome of pulmonary rehabilitation in COPD. Respir Med. 2001 Jan;95(1):71-7. doi: 10.1053/rmed.2000.0976. PMID 11207021
- [Background] Revill SM, Morgan MD, Singh SJ, Williams J, Hardman AE. The endurance shuttle walk: a new field test for the assessment of endurance capacity in chronic obstructive pulmonary disease. Thorax. 1999 Mar;54(3):213-22. doi: 10.1136/thx.54.3.213. PMID 10325896
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Singh SJ, Morgan MD, Hardman AE, Rowe C, Bardsley PA. Comparison of oxygen uptake during a conventional treadmill test and the shuttle walking test in chronic airflow limitation. Eur Respir J. 1994 Nov;7(11):2016-20. PMID 7875275
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Eaton T, Young P, Nicol K, Kolbe J. The endurance shuttle walking test: a responsive measure in pulmonary rehabilitation for COPD patients. Chron Respir Dis. 2006;3(1):3-9. doi: 10.1191/1479972306cd077oa. PMID 16509172
- [Background] Ozcan A, Donat H, Gelecek N, Ozdirenc M, Karadibak D. The relationship between risk factors for falling and the quality of life in older adults. BMC Public Health. 2005 Aug 26;5:90. doi: 10.1186/1471-2458-5-90. PMID 16124871
- [Background] Steiner MC, Barton RL, Singh SJ, Morgan MD. Bedside methods versus dual energy X-ray absorptiometry for body composition measurement in COPD. Eur Respir J. 2002 Apr;19(4):626-31. doi: 10.1183/09031936.02.00279602. PMID 11998990
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Garrod R, Ansley P, Canavan J, Jewell A. Exercise and the inflammatory response in chronic obstructive pulmonary disease (COPD)--Does training confer anti-inflammatory properties in COPD? Med Hypotheses. 2007;68(2):291-8. doi: 10.1016/j.mehy.2006.07.028. Epub 2006 Sep 28. PMID 17010529
- [Background] O'Neill B, McKevitt A, Rafferty S, Bradley JM, Johnston D, Bradbury I, McMahon J. A comparison of twice- versus once-weekly supervision during pulmonary rehabilitation in chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2007 Feb;88(2):167-72. doi: 10.1016/j.apmr.2006.11.007. PMID 17270513
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Derived] Wilson AM, Browne P, Olive S, Clark A, Galey P, Dix E, Woodhouse H, Robinson S, Wilson EC, Staunton L. The effects of maintenance schedules following pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a randomised controlled trial. BMJ Open. 2015 Mar 11;5(3):e005921. doi: 10.1136/bmjopen-2014-005921. PMID 25762226